CLINICAL TRIAL: NCT00437931
Title: Color Flow Doppler Ultrasound in Subclinical Thyroid Dysfunction
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, avraham ishay, Dr, HaEmek Medical Center, Israel
Other Study IDs: 006-07-EMC
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Subclinical Hypothyroidism; Hyperthyroidism; Thyroid Dysfunction
Keywords: hypothyroidism; hyperthyroidism; thyroid dysfunction; ultrasound; doppler
MeSH Terms: conditions — Hyperthyroidism; Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- A: patients with subclinical hypothyroidism
- B: patients with subclinical hyperthyroidism
- C: patient with normal thyroid function.

SUMMARY:
Overt hyperthyroidism and hypothyroidism are associated with inverted hemodynamic changes.Regional blood flow disturbances (including intrathyroidal) were also reported in these thyroid disorders. The purpose of this study is to investigate the thyroid vascularity and blood flow by Color Flow Doppler Sonography in patients with subclinical thyroid dysfunction

DETAILED DESCRIPTION:
Color Flow Doppler Sonography (CFDS) has become in the last years an increasing procedure to assess the thyroid blood flow. Previous studies showed specific changes of thyroid blood flow in hyperthyroidism, Hashimoto's thyroiditis and thyroid nodules when investigated by CFDS. Subclinical hyperthyroidism and hypothyroidism are common laboratory findings, defined by normal thyroid hormones concentrations along with ,respectively,decreased or increase Thyroid stimulating hormone (TSH) level. We purpose to investigate thyroid vascularity by CFDS in patients with subclinical hyperthyroidism or hypothyroidism and compared them with euthyroid patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with subclinical hypothyroidism or hyperthyroidism
* patients with thyroid nodules and normal thyroid function

Exclusion Criteria:

* patients who are taking thyroxine, antithyroid drugs, lithium or amiodarone
* patients who had thyroid surgery or radioiodine therapy
* patients with NYHA class 3 or 4 heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with subclinical hypothyroidism and hyperthyroidism
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Ishay, MD, Principal Investigator — Haemek Medical Center, Endocrine Institute, Afula, Israel; Leonid Chervinsky, Study Chair — Haemek Medical Center, Department of Radiology, Afula , Israel; Rafael Luboshitzky, MD, Study Chair — Haemek Medical Center, Endocrine Institute, Afula, Israel
Locations (1):
- Haemek Medical Center, Department of Radiology, Afula, Israel